CLINICAL TRIAL: NCT00954317
Title: Do Epidurals Placed at a Lower Level Improve Labour Analgesia
Brief Title: Do Epidurals Placed at a Lower Level Improve Labor Analgesia?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Victoria Hospital, Canada (Other)
Responsible Party: Principal Investigator, Albert Moore, Dr., Royal Victoria Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDR-08-052
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Labor Analgesia
Keywords: epidural; labour analgesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low epidural (Active Comparator): epidural placed in the lower lumbar vertebral column
  Interventions: Procedure: epidural placed low
- high epidural (Experimental): high epidural
  Interventions: Procedure: high epidural

INTERVENTIONS:
Procedure: epidural placed low — epidural placed low
  Arms: Low epidural
Procedure: high epidural — high epidural
  Arms: high epidural

SUMMARY:
The investigators wish to compare the analgesia provided by epidurals placed high in the lumbar spine versus epidurals place low in the lumbar spine.

ELIGIBILITY:
Inclusion Criteria:

* women in active labor

Exclusion Criteria:

* known contraindications to epidural analgesia
* moderate to severe systemic illness as evidenced by an American Society of Anesthesiologists (ASA) score of 3 or higher.
* known abnormalities of the spinal column
* any neurologic illness
* multiple gestations, fetal abnormalities or fetal presentation other than vertex
* recent history of analgesic usage
* an inability to communicate in English or French
* Body Mass Index greater than 40
* patients in pain requesting an immediate epidural

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Number of epidural medication boluses required | 30 minutes and 1 hour

SECONDARY OUTCOMES:
Labour progress | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Moore A, Villeneuve V, Bravim B, El-Bahrawy A, El-Mouallem E, Kaufman I, Hatzakorzian R, Li Pi Shan W. The Labor Analgesia Requirements in Nulliparous Women Randomized to Epidural Catheter Placement in a High or Low Intervertebral Space. Anesth Analg. 2017 Dec;125(6):1969-1974. doi: 10.1213/ANE.0000000000002076. PMID 28504988